CLINICAL TRIAL: NCT06526650
Title: The PILI 'Āina Project
Brief Title: 'Ai Pono Cooking Demonstrations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: National Institutes of Health (NIH) (NIH); American Heart Association (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PILI 'Āina 3; R01HL168858 (NIH)
Record Dates: First submitted 2024-06-07; First posted 2024-07-30 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes; Hypertension; Dyslipidemias; Overweight and Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Dyslipidemias; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Aim 3: Community Level Intervention (Other): Aim 3 is community-driven, supports the overall goal of the PILI 'Āina project, allows all members of the community to benefit, and is strongly promoted within the community. The investigators will design and implement 'Ai Pono, a community-level component that can operate in tandem with PILI 'Āina. This component will not be tested in the group-randomized trial. Instead, all 7 communities will implement 'Ai Pono for the full study period.
  Interventions: Other: 'Ai Pono

INTERVENTIONS:
Other: 'Ai Pono — "Hands-on Cooking and Cultural Lessons" These lessons will be widely advertised. Each 2-hour presentation will involve hands-on cooking demonstrations and tastings, accompanied by lessons on the cultural significance of featured food items. Demonstrations will link the consumption of vegetables (e.g., sweet potato, breadfruit, kalo) to Native Hawaiian (NH) history and traditional beliefs to help participants rediscover their heritage through the meals they prepare.

SUMMARY:
Native Hawaiians' traditional lifestyles and diets ensured the mutual health and well-being of the land and its inhabitants, which stand in stark contrast to the disproportionately high prevalence of diet-related, cardiometabolic diseases they experience today. In this project, the investigators will adapt and test an evidence-based multilevel intervention entitled PILI 'Āina to improve the self-management of prevalent cardiometabolic diseases and reduce risk factors for developing new diet-related illnesses and implement and evaluate the impact and sustainability of community-wide cooking demonstrations. The objectives of this project are to optimize the effectiveness and sustainability of PILI 'Āina, improve diet quality, cardiometabolic markers, promote traditional Native Hawaiian diets, and improve social cohesion.

DETAILED DESCRIPTION:
In Years 1 - 5, the investigators will hold quarterly cooking demonstrations and cultural lessons for a total of 36 events. The lessons will be aimed at improving family and community eating environments of participants and social cohesion of these communities. Attendance at each lesson will be limited to 30 individuals. Attendees will register via REDCap using their names and email addresses. There is no limit to how many lessons an individual can attend, but after the first lesson the investigators reserve 15 of the 30 spots for people who have not attended previously, as identified by their registration information. At each quarterly event, the investigators survey participants to assess their reaction to the lesson, their vegetable and fruit intake, self-efficacy for healthy diet, and perceptions of community cohesion. Surveys will take ~5-10 minutes to complete. Additionally, the investigators will survey random samples of homestead households (n = 20 per homestead, total n = 140 per year) in Projects Years 1 - 5. Total sample for this activity is 700. Each sample will be selected independent of previous samples, and it is possible the same households will be sampled multiple times.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ (looking for older adults)
* Native Hawaiian resident in a participating homestead
* Overweight or obese (BMI ≥ 25 kg/m^2)
* Prior diagnosis of type 2 diabetes or pre-diabetes, hypertension, and/or dyslipidemia (LDL cholesterol ≥ 130 mg/dL)
* Capable of 150 minutes of moderate physical activity (e.g., brisk walking) per week
* Willing and able to participate in all aspects of the individual and household-level intervention
* Fluent in written and spoken English

Exclusion Criteria:

* No children
* Pregnancy
* Serious illness such as cancer or chronic pain that may contraindicate full participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1780 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2028-03-06 (Estimated); Study Completion 2028-03-13 (Estimated)

PRIMARY OUTCOMES:
Family Environment | Baseline, 1-year, 2-year, 3-year, 4-year
  Three subscales, Cohesion, Expressiveness, and Conflict, assess the degree of commitment and support family members provide for one another, the extent to which family members are encouraged to express their feelings directly, and the amount of openly expressed anger and conflict among family members.
Nutrition Environment | Baseline, 1-year, 2-year, 3-year, 4-year
  The perceived 9-item nutrition environment will be measured by the Gustafson Perceived Nutrition Environment Measures questionnaire, which examines perceived access and availability of healthy foods within ~1 mile of the participant's home, and the availability and affordability of produce in the participant's primary food store. The responses and scores vary depending on the question including 0- disagree, 1-agree, and 0-not important, 1-slightly important, 2-moderately important, 3- important, 4-very important. Higher scores indicate higher perceived access and availability of food.
Social Cohesionn | Baseline, 1-year, 2-year, 3-year, 4-year
  4-item subscale of the neighborhood level stressors which asks about perceived shared values and trust.

SECONDARY OUTCOMES:
Diet Self-Efficacy | Baseline, 1-year, 2-year, 3-year, 4-year
  The 11-item Diet Self Efficacy Scale will measure self-efficacy in avoiding tempting high caloric food and managing social and internal cues and negative emotions. The responses and scores range from 1-strongly disagree, 2-somewhat disagree, 3-neutral, 4-somewhat agree, and 5-strongly agree. Higher scores indicate greater self-efficacy with diet.
Food Literacy | Baseline, 1-year, 2-year, 3-year, 4-year
  Food literacy, defined as the ability to make healthy food choices in different settings and situations, will be assessed by the 11-item self-perceived food literacy scale, which encompasses knowledge, skills, and behaviors pertinent to planning, selecting, preparing, and eating healthy food. The responses and scores range from 1-not at all/never, 2-disagree, 3-slightly disagree, 4- slightly agree, 5-yes/always. Higher scores indicate greater food literacy.
Social Support | Baseline, 1-year, 2-year, 3-year, 4-year
  Social support for a healthy diet will be measured as the perceived support that people who make dietary changes receive from family and friends. An 11-item questionnaire on social support will be used to ask participants' perceived level of support from friends and family regarding diet choices. The responses and scores range from 1-strongly disagree, 2-somewhat disagree, 3-neutral, 4-somewhat agree, and 5-strongly agree. Higher scores indicate greater social support.

OTHER OUTCOMES:
Cultural Identity | Baseline, 1-year, 2-year, 3-year, 4-year
  Cultural factors will be measured by the 4-item Cultural Identity Scale that will assess the degree of identification with NH cultural heritage. The responses and scores range from 0-not at all knowledgeable, 1- somewhat not knowledgeable, 2-neutral or no response, 3-somewhat knowledgeable, and 4-very knowledgeable. Higher scores indicate greater cultural identity.
Demographic Data- Date of Birth | Baseline, 1-year, 2-year, 3-year, 4-year
  Date of birth:
  * Month
  * Day
  * Year
Demographic Data- Biological Sex | Baseline, 1-year, 2-year, 3-year, 4-year
  Biological Sex:
  * Female
  * Male
Demographic Data- Marital status | Baseline, 1-year, 2-year, 3-year, 4-year
  Marital Status:
  * Never married
  * Currently married
  * Divorced or separated
  * Widow/widower
  * Domestic partnership/other
Demographic Data- Employment | Baseline, 1-year, 2-year, 3-year, 4-year
  Employment:
  * Full time
  * Part-time
  * Unemployed
  * Self-employed
  * Retired
  * Unable to work/other
  * Household caretaker
Demographic Data- Education | Baseline, 1-year, 2-year, 3-year, 4-year
  Education:
  * Less than high school
  * High school diploma/General Education Diploma (GED)
  * Some college/technical training
  * College degree
  * Graduate/professional degree
Demographic Data- Ethnic ancestry | Baseline, 1-year, 2-year, 3-year, 4-year
  Ethnic Ancestry:
  * Caucasian
  * Chinese
  * Filipino
  * Hawaiian
  * Latino
  * Japanese
  * Korean
  * Marshallese
  * Micronesian (specify)
  * Native American
  * Portuguese
  * Samoan
  * Other (specify)
Demographic Data- Household income | Baseline, 1-year, 2-year, 3-year, 4-year
  Household Income:
  * Under $49,999
  * $50,000-$74,999
  * $75,000-$99,999
  * $100,000-$124,999
  * Over $125,000
  Household income will be classified according to the US Census Bureau's poverty threshold by using a dichotomous variable. Participation in public assistance programs (e.g., Temporary Assistance for Needy Families, Supplemental Nutrition Assistance Program) will also be recorded.
Demographic Data- Household Composition | Baseline, 1-year, 2-year, 3-year, 4-year
  Household Composition:
  1. Who lives in the participant's house full-time? (50% or more time spent in-house)
  * Parents
  * Children
  * Grandparents/great-grandparents
  * Other family members
    a. Of those people, what are their ages and genders?
  * Male: 17 years and under, 18-29 yrs, 30-39 yrs, 40-39 yrs, 50-59 yrs, 60+ yrs
  * Female: 17 years and under, 18-29 yrs, 30-39 yrs, 40-39 yrs, 50-59 yrs, 60+ yrs
  * Number of other/non-binary: 17 years and under, 18-29 yrs, 30-39 yrs, 40-39 yrs, 50-59 yrs, 60+ yrs

CONTACTS AND LOCATIONS:
Overall Officials: Claire Ing, DrPH, Principal Investigator — Principal Investigator; Kulani DeSimone, B.S., Study Chair — Graduate Assistant
Locations (2):
- United States (2):
  - Kula no na Poe Hawaii, Honolulu, Hawaii
  - Kapolei Community Development Coalition, Kapolei, Hawaii